CLINICAL TRIAL: NCT02021526
Title: Treatment Development of Triheptanoin for Glucose Transporter Type I Deficiency
Brief Title: Triheptanoin (C7 Oil), a Food Supplement, for Glucose Transporter Type I Deficiency (G1D)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: NIH funding resulted in new clinical trial
Sponsor: Juan Pascual (Other)
Responsible Party: Sponsor-Investigator, Juan Pascual, Associate Professor, Director of the Rare Brain Disorders Program, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PASCG1D2014
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome; Glut1 Deficiency Syndrome
Keywords: G1D; Glut1 Deficiency; Glucose Transporter Type 1 Deficiency; Glucose Transporter Type I Deficiency
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Dietary Therapy (Experimental): Patients currently on no dietary therapy will receive triheptanoin (C7 oil), dosed at 1 g/kg body weight and divided into 4 doses daily, administered for 6 months
  Interventions: Drug: Triheptanoin
- Ketogenic Diet (Experimental): Patients on ketogenic diet will receive triheptanoin (C7 oil) in place of their usual fat intake, at a dose sufficient to maintain their ketogenic diet ratio (based on patient weight and current ratio). Patients will receive triheptanoin for 6 months.
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Triheptanoin (C7 oil) is a 7-carbon medium chain triglyceride.
  Other Names: C7; Heptanoate; Heptanoic Acid

SUMMARY:
This is a single-site, open-label, phase II trial of C7, a food supplement or medical food, for the development of treatment outcome measures for glucose transporter type I deficiency (G1D). The primary outcome measures are: 1. Safety and tolerability of C7 as measured by changes in comprehensive blood work, including lipid and free fatty acid panels, self-reported side effects and clinical exam; 2. Changes in brain metabolic rate by MRI and EEG measurements during C7 treatment; and 3. Maintenance of ketosis in G1D patients on ketogenic diet, as measured by serial ketone levels during treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or suspected diagnosis of glucose transporter type I deficiency (G1D).
* On stable ketogenic diet at a ratio between 1:2.5 and 1:4 OR Stable on no dietary therapy
* Males and females 30 months to 55 years old, inclusive.

Exclusion Criteria:

* Subjects with a history of life-threatening seizure episodes, including but not limited to status epilepticus and cardiac arrest.
* Subjects with a BMI (body mass index) greater than or equal to 30 will be excluded.
* Subjects currently on dietary therapy other than ketogenic diet (i.e., medium chain triglyceride-supplemented diets, Atkins diet, low glycemic index diet, etc.).
* Women who are pregnant or breast-feeding may not participate. Women who plan to become pregnant during the course of the study, or who are unwilling to use birth control to prevent pregnancy (including abstinence) may not participate.
* Allergy/sensitivity to triheptanoin.
* Previous treatment with triheptanoin.
* Treatment with medium chain triglycerides in the last 30 days.
* Subjects exhibiting signs of dementia, or diagnosed with any degenerative brain disorder (such as Alzheimer's disease) that would confound assessment of cognitive changes, in the opinion of the investigator.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Patients with metal implants, experience claustrophobia, or who are behaviorally unable to be still for MRS (magnetic resonance spectroscopy) imaging (not due to seizures) will be excluded from the imaging portion of the research.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent, or assent for children age 10-17.

Ages: 30 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in risk for Metabolic Syndrome | Baseline, 6 months, 9 months
  Triglycerides, lipid levels, and cholesterol are measured to evaluate change in risk of metabolic syndrome
Change on Biomarkers | Baseline, 6 months, 9 months
  EEG and brain metabolic rate will be measured at three time points. Changes in these biomarkers indicate the utilization of triheptanoin in brain metabolism
Change in Ketosis | baseline, 6 months, 9 months
  Safety blood work (described in the first outcome measure) is measured along with ketone levels and EEG to confirm that triheptanoin is safe and does not break ketosis in patients on the ketogenic diet

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pascual, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Marin-Valencia I, Good LB, Ma Q, Duarte J, Bottiglieri T, Sinton CM, Heilig CW, Pascual JM. Glut1 deficiency (G1D): epilepsy and metabolic dysfunction in a mouse model of the most common human phenotype. Neurobiol Dis. 2012 Oct;48(1):92-101. doi: 10.1016/j.nbd.2012.04.011. Epub 2012 Apr 23. PMID 22683290
- [Background] Jeffrey FM, Marin-Valencia I, Good LB, Shestov AA, Henry PG, Pascual JM, Malloy CR. Modeling of brain metabolism and pyruvate compartmentation using (13)C NMR in vivo: caution required. J Cereb Blood Flow Metab. 2013 Aug;33(8):1160-7. doi: 10.1038/jcbfm.2013.67. Epub 2013 May 8. PMID 23652627
- [Background] Xu F, Liu P, Pascual JM, Xiao G, Lu H. Effect of hypoxia and hyperoxia on cerebral blood flow, blood oxygenation, and oxidative metabolism. J Cereb Blood Flow Metab. 2012 Oct;32(10):1909-18. doi: 10.1038/jcbfm.2012.93. Epub 2012 Jun 27. PMID 22739621
- [Background] Marin-Valencia I, Good LB, Ma Q, Jeffrey FM, Malloy CR, Pascual JM. High-resolution detection of (1)(3)C multiplets from the conscious mouse brain by ex vivo NMR spectroscopy. J Neurosci Methods. 2012 Jan 15;203(1):50-5. doi: 10.1016/j.jneumeth.2011.09.006. Epub 2011 Sep 17. PMID 21946227
- [Background] Marin-Valencia I, Roe CR, Pascual JM. Pyruvate carboxylase deficiency: mechanisms, mimics and anaplerosis. Mol Genet Metab. 2010 Sep;101(1):9-17. doi: 10.1016/j.ymgme.2010.05.004. Epub 2010 Jun 9. PMID 20598931
- [Background] Perez-Duenas B, Prior C, Ma Q, Fernandez-Alvarez E, Setoain X, Artuch R, Pascual JM. Childhood chorea with cerebral hypotrophy: a treatable GLUT1 energy failure syndrome. Arch Neurol. 2009 Nov;66(11):1410-4. doi: 10.1001/archneurol.2009.236. PMID 19901175
- [Background] Pascual JM, Campistol J, Gil-Nagel A. Epilepsy in inherited metabolic disorders. Neurologist. 2008 Nov;14(6 Suppl 1):S2-S14. doi: 10.1097/01.nrl.0000340787.30542.41. PMID 19225367
- [Background] Pascual JM, Wang D, Lecumberri B, Yang H, Mao X, Yang R, De Vivo DC. GLUT1 deficiency and other glucose transporter diseases. Eur J Endocrinol. 2004 May;150(5):627-33. doi: 10.1530/eje.0.1500627. PMID 15132717
- [Background] Pascual JM, Wang D, Yang R, Shi L, Yang H, De Vivo DC. Structural signatures and membrane helix 4 in GLUT1: inferences from human blood-brain glucose transport mutants. J Biol Chem. 2008 Jun 13;283(24):16732-42. doi: 10.1074/jbc.M801403200. Epub 2008 Apr 3. PMID 18387950
- [Background] Pascual JM, Wang D, Hinton V, Engelstad K, Saxena CM, Van Heertum RL, De Vivo DC. Brain glucose supply and the syndrome of infantile neuroglycopenia. Arch Neurol. 2007 Apr;64(4):507-13. doi: 10.1001/archneur.64.4.noc60165. Epub 2007 Feb 12. PMID 17296829
- [Background] Pascual JM. [Glucose transport hereditary diseases]. Med Clin (Barc). 2006 Nov 11;127(18):709-14. doi: 10.1157/13095099. Spanish. PMID 17169300
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Mao X, Cheng J, Yoo J, Noebels JL, De Vivo DC. A mouse model for Glut-1 haploinsufficiency. Hum Mol Genet. 2006 Apr 1;15(7):1169-79. doi: 10.1093/hmg/ddl032. Epub 2006 Feb 23. PMID 16497725
- [Background] Wang D, Pascual JM, Yang H, Engelstad K, Jhung S, Sun RP, De Vivo DC. Glut-1 deficiency syndrome: clinical, genetic, and therapeutic aspects. Ann Neurol. 2005 Jan;57(1):111-8. doi: 10.1002/ana.20331. PMID 15622525
- [Background] Pascual JM, Lecumberri B, Wang D, Yang R, Engelstad K, De Vivo DC. [Type 1 glucose transporter (Glut1) deficiency: manifestations of a hereditary neurological syndrome]. Rev Neurol. 2004 May 1-15;38(9):860-4. Spanish. PMID 15152356
- [Background] Wang D, Pascual JM, Iserovich P, Yang H, Ma L, Kuang K, Zuniga FA, Sun RP, Swaroop KM, Fischbarg J, De Vivo DC. Functional studies of threonine 310 mutations in Glut1: T310I is pathogenic, causing Glut1 deficiency. J Biol Chem. 2003 Dec 5;278(49):49015-21. doi: 10.1074/jbc.M308765200. Epub 2003 Sep 16. PMID 13129919
- [Background] Pascual JM, Van Heertum RL, Wang D, Engelstad K, De Vivo DC. Imaging the metabolic footprint of Glut1 deficiency on the brain. Ann Neurol. 2002 Oct;52(4):458-64. doi: 10.1002/ana.10311. PMID 12325075
- [Background] Iserovich P, Wang D, Ma L, Yang H, Zuniga FA, Pascual JM, Kuang K, De Vivo DC, Fischbarg J. Changes in glucose transport and water permeability resulting from the T310I pathogenic mutation in Glut1 are consistent with two transport channels per monomer. J Biol Chem. 2002 Aug 23;277(34):30991-7. doi: 10.1074/jbc.M202763200. Epub 2002 May 24. PMID 12032147
- [Background] De Vivo DC, Wang D, Pascual JM, Ho YY. Glucose transporter protein syndromes. Int Rev Neurobiol. 2002;51:259-88. doi: 10.1016/s0074-7742(02)51008-4. No abstract available. PMID 12420362
- [Background] Brockmann K, Wang D, Korenke CG, von Moers A, Ho YY, Pascual JM, Kuang K, Yang H, Ma L, Kranz-Eble P, Fischbarg J, Hanefeld F, De Vivo DC. Autosomal dominant glut-1 deficiency syndrome and familial epilepsy. Ann Neurol. 2001 Oct;50(4):476-85. doi: 10.1002/ana.1222. PMID 11603379
- [Background] Marin-Valencia I, Yang C, Mashimo T, Cho S, Baek H, Yang XL, Rajagopalan KN, Maddie M, Vemireddy V, Zhao Z, Cai L, Good L, Tu BP, Hatanpaa KJ, Mickey BE, Mates JM, Pascual JM, Maher EA, Malloy CR, Deberardinis RJ, Bachoo RM. Analysis of tumor metabolism reveals mitochondrial glucose oxidation in genetically diverse human glioblastomas in the mouse brain in vivo. Cell Metab. 2012 Jun 6;15(6):827-37. doi: 10.1016/j.cmet.2012.05.001. PMID 22682223
- [Background] Maher EA, Marin-Valencia I, Bachoo RM, Mashimo T, Raisanen J, Hatanpaa KJ, Jindal A, Jeffrey FM, Choi C, Madden C, Mathews D, Pascual JM, Mickey BE, Malloy CR, DeBerardinis RJ. Metabolism of [U-13 C]glucose in human brain tumors in vivo. NMR Biomed. 2012 Nov;25(11):1234-44. doi: 10.1002/nbm.2794. Epub 2012 Mar 15. PMID 22419606
- [Background] Marin-Valencia I, Cho SK, Rakheja D, Hatanpaa KJ, Kapur P, Mashimo T, Jindal A, Vemireddy V, Good LB, Raisanen J, Sun X, Mickey B, Choi C, Takahashi M, Togao O, Pascual JM, Deberardinis RJ, Maher EA, Malloy CR, Bachoo RM. Glucose metabolism via the pentose phosphate pathway, glycolysis and Krebs cycle in an orthotopic mouse model of human brain tumors. NMR Biomed. 2012 Oct;25(10):1177-86. doi: 10.1002/nbm.2787. Epub 2012 Mar 1. PMID 22383401
- [Background] Choi C, Ganji SK, DeBerardinis RJ, Hatanpaa KJ, Rakheja D, Kovacs Z, Yang XL, Mashimo T, Raisanen JM, Marin-Valencia I, Pascual JM, Madden CJ, Mickey BE, Malloy CR, Bachoo RM, Maher EA. 2-hydroxyglutarate detection by magnetic resonance spectroscopy in IDH-mutated patients with gliomas. Nat Med. 2012 Jan 26;18(4):624-9. doi: 10.1038/nm.2682. PMID 22281806
- [Background] Choi C, Ganji SK, DeBerardinis RJ, Dimitrov IE, Pascual JM, Bachoo R, Mickey BE, Malloy CR, Maher EA. Measurement of glycine in the human brain in vivo by 1H-MRS at 3 T: application in brain tumors. Magn Reson Med. 2011 Sep;66(3):609-18. doi: 10.1002/mrm.22857. Epub 2011 Mar 9. PMID 21394775